CLINICAL TRIAL: NCT03037255
Title: Association of Long-term Conditions With Survival Following Acute Myocardial Infarction in England and Wales
Brief Title: Association of Long-term Conditions With Survival Following Heart Attack in England and Wales
Status: Completed | Type: Observational
Sponsor: Marlous Hall (Other)
Responsible Party: Sponsor-Investigator, Marlous Hall, Co-Investigator, University of Leeds
Organization: University of Leeds (Other)
Other Study IDs: UoL_LTC
Record Dates: First submitted 2017-01-24; First posted 2017-01-31 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Acute Myocardial Infarction; Diabetes Mellitus; Peripheral Vascular Disease; Chronic Heart Failure; Cerebrovascular Disease; Chronic Renal Failure; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Vascular Diseases; Cerebrovascular Disorders; Kidney Failure, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: long term conditions — Long term conditions including diabetes mellitus, chronic obstructive pulmonary disease or asthma, chronic heart failure, chronic renal failure, cerebrovascular disease or peripheral vascular disease.

SUMMARY:
This study aims to determine the extent to which pre-existing long-term conditions are associated with survival following a heart attack (acute myocardial infarction) using observational data from the UK's national heart attack register.

DETAILED DESCRIPTION:
Using observational data from the Myocardial Ischaemia National Audit Project (MINAP) of all hospitalisations for acute myocardial infarction in all acute hospitals in England and Wales, this study aims to determine the extent to which pre-existing long-term conditions are associated with survival following acute myocardial infarction. The study will include an investigation of individual long term conditions for patients with acute myocardial infarction, including chronic heart failure, cerebrovascular disease, diabetes mellitus, chronic obstructive pulmonary disease, chronic renal failure or peripheral vascular disease as well as the combination of such conditions and their resulting impact on long term all-cause mortality (up to 8.4 years). In addition, an investigation of the association of receipt of guideline recommended care for acute myocardial infarction patients with pre-existing long term conditions will be made.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older

Exclusion Criteria:

* Patients for which mortality data are missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ST-segment elevation myocardial infarction (STEMI) or non-STEMI (NSTEMI) admitted to one of 247 hospitals in England and Wales between 1st January 2003 and 30th June 2013
Sampling Method: Non-Probability Sample
Enrollment: 693633 (Actual)
Dates: Start 2003-01; Primary Completion 2013-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who died from any cause by the end of the study censoring period | 8.4 years
  Death data was obtained from national death records from the Office for National Statistics

SECONDARY OUTCOMES:
Number of patients who received guideline recommended therapy during the study period | Any guideline therapy administered during the patients hospital admission for acute myocardial infarction, an average of 4 days
  All guideline recommended therapies for acute myocardial infarction relevant to the duration of the study period (2003 to 2013) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Gale, PhD, FRCP, Principal Investigator — University of Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall M, Dondo TB, Yan AT, Mamas MA, Timmis AD, Deanfield JE, Jernberg T, Hemingway H, Fox KAA, Gale CP. Multimorbidity and survival for patients with acute myocardial infarction in England and Wales: Latent class analysis of a nationwide population-based cohort. PLoS Med. 2018 Mar 6;15(3):e1002501. doi: 10.1371/journal.pmed.1002501. eCollection 2018 Mar. PMID 29509764
- See also: Principal Researchers Profile Page — https://medicinehealth.leeds.ac.uk/medicine/staff/390/dr-marlous-hall